CLINICAL TRIAL: NCT06133504
Title: Association Between Early Multimodal Therapy and Mechanical Ventilation Days in the Intensive Care Unit at Fundación Santa Fe de Bogotá: A Randomized Controlled Clinical Trial
Brief Title: Early Multimodal Therapy and Mechanical Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Jorge Iván Alvarado, Principal investigator, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SECEC-2023-129
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Critical Care; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: The study is a phase III randomized clinical trial at a single center with two patient groups, "early arm" (EA) and "late arm," assigned through stratified randomization. Allocation concealment uses sealed envelopes. EA includes intubated patients receiving early multimodal therapy, while the "late arm" starts therapy during ventilatory support weaning. Blinding isn't feasible, but final assessments at 90 days are blinded to intervention groups. Statisticians analyze data blinded. The study is intention-to-treat based, ensuring a comprehensive evaluation of intervention effectiveness
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early arm (Active Comparator): Early multimodal therapy is characterized by a comprehensive set of therapeutic interventions executed by the physiotherapy, speech therapy, respiratory therapy, and occupational therapy teams precisely at the moment of study inclusion. This tailored approach ensures that patients receive a coordinated and multidisciplinary therapeutic regimen right from the outset of their participation in the study
  Interventions: Procedure: Early Multimodal Therapy
- Late arm (Active Comparator): While late multimodal therapy is characterized by the same type of maneuvers carried out by the same disciplinary team but initiated once indicated by the attending physician.
  Interventions: Procedure: Late Multimodal Therapy

INTERVENTIONS:
Procedure: Early Multimodal Therapy — Early multimodal therapy is defined as the collection of therapeutic maneuvers performed by the physiotherapy, speech therapy, respiratory therapy, and occupational therapy team at the time of study inclusion.
  Arms: Early arm
Procedure: Late Multimodal Therapy — Late multimodal therapy is characterized by the same set of maneuvers carried out by the same disciplinary team, but it is initiated once indicated by the attending physician.
  Arms: Late arm

SUMMARY:
To assess the association between early multimodal therapy and the duration of invasive mechanical ventilation in the Intensive Care Unit at Fundación Santa Fe de Bogotá.

DETAILED DESCRIPTION:
This study compares the impact of early multimodal therapy on mechanical ventilation duration in ICU patients. It is an open-label, randomized controlled clinical trial. Patients will be assigned to either early multimodal therapy or standard therapy (control) in a 1:1 ratio. Blinding is not possible due to the study design. The analysis will follow an intention-to-treat approach. The hypothesis is that early multimodal therapy reduces mechanical ventilation duration

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are as follows:

Patients hospitalized in the adult intensive care unit of the Fundación Santa Fe de Bogotá.

Requirement of invasive mechanical ventilation through an endotracheal tube for a period exceeding 72 hours with an expected continuation of at least 24 hours.

Barthel Index equal to or greater than 70

Exclusion Criteria:

* Invasive mechanical ventilation through tracheostomy or a nasotracheal tube.
* History of head and neck surgery at any time prior to ICU admission.
* Patients directly admitted to the ICU due to cardiac arrest by any cause.
* Airway burn.
* Burns involving ≥ 50% of the body surface area.
* Chronic obstructive pulmonary disease (these patients usually require prolonged mechanical ventilation due to the underlying respiratory dysfunction)
* Patients referred from another institution.
* Demyelinating diseases or neuromuscular junction disorders at ICU admission.
* Patients requiring neuromuscular blockade.
* Patients with a life expectancy of ≤180 days will be excluded based on their primary diagnosis (e.g., advanced cancer, end-stage heart failure), comorbidities, recent clinical course, medical judgment by the ICU team, and functional status as assessed by the Barthel index.
* ICU readmissions.
* Participation in other rehabilitation clinical trials.
* Liver or kidney transplant.
* Patients with an active cancer diagnosis undergoing oncological treatment (chemotherapy/surgery) at the time of eligibil- ity assessment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time (days) from intubation to extubation. | 28 days
  Days of mechanical ventilation duration

SECONDARY OUTCOMES:
Ventilator-free days until day 28 | 28 days
  28 minus the days of mechanical ventilation
Delirium days until day 28 | 28 days
  In order for a patient to be considered to have delirium according to the CAM-ICU, the first criterion (acute change in mental status) must be present, along with at least one of the other three criteria (inability to maintain sustained attention, disorganized thinking, or fluctuating levels of consciousness).
Delirium-free days until day 28 | 28 days
  28 minus days with presence of delirium
Sedation days until day 28. | 28 days
  Sedation days until day 28.
Sedation-free days until day 28 | 28 days
  28 days minus days of sedation
Barthel Index at hospital discharge | 28 days
  The Barthel Index is a scale used to measure the degree of functional independence in activities of daily living (ADLs) for an individual. The score is 0 if the patient deceases.
Hospitalization days | 90 days
  Hospitalization days
ICU length of stay | 28 days
  ICU length of stay
Mortality from any cause up to 90 days | 90 days
  Mortality from any cause up to 90 days
Functional independence status measured by ADLs at hospital discharge | 90 days
  Activities of Daily Living (ADLs), each variable scores one point: bathing, dressing, eating, grooming, transferring from bed to chair, and using the bathroom
Functional independence status measured by ADLs at ICU discharge | 28 days
  Activities of Daily Living (ADLs), each variable scores one point: bathing, dressing, eating, grooming, transferring from bed to chair, and using the bathroom
Muscle strength measured using the Medical Research Council (MRC) scale | 28 days
  Muscle strength assessment in critical care patients using the Medical Research Council (MRC) scale:
  5: Normal - Full range of motion against total resistance 4+: Good (+) - Full range of motion against gravity and strong resistance 4: Good (-) - Full range of motion against gravity and minimal resistance 3+: Fair (+) - Full range of motion against gravity only 3: Fair (-) - Partial range of motion against gravity 2: Poor - Movement with gravity eliminated
  1: Minimal - Visible muscle contraction without movement 0: Absent - Total paralysis
Swallowing difficulty at 72 hours. | 28 days
  Presence of dysphagia at 72 hours after extubation
Time until the initiation of oral intake | 28 days
  Time to initiate oral intake after extubation: 1) 12-24 hours, 2) > 24 hours
Development of healthcare-associated pneumonia | 28 days
  Pneumonia associated with invasive mechanical ventilation. Yes or no.
Maximum mobility measured by JH-HLM (Johns Hopkins Highest Level of Mobility) scale | 28 days
  Mobility assessment using the JH-HLM (Johns Hopkins Highest Level of Mobility) scale:
  8: Walks more than 250 feet. 7: Walks more than 25 feet. 6: Walks more than 10 steps. 5: Stands for more than one minute. 4: Can move to the chair. 3: Can sit on the edge of the bed. 2: Can turn in bed.
  1: Can only lie down. Score is 0 if the patient deceases.
Grip strength | 28 days
  Grip strength of the dominant hand within 24 hours post-extubation. Kilograms. Score is 0 if the patient deceases
Extubation failure | 28 days
  Inability to breathe spontaneously in the first 48 hours after removal of artificial airway, and the patient is unable to maintain a patent airway
Need for non-invasive mechanical ventilation | 28 days
  Need for non-invasive mechanical ventilation: Yes or No
Cognitive function measured using the Montreal Cognitive Assessment (MOCA). | 90 days
  The variable is the cognitive function, assessed using the Montreal Cognitive Assessment (MOCA). This tool measures various cognitive domains, providing insight into an individual's cognitive abilities and identifying potential cognitive impairment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarado Sanchez JI, Castillo Morales LM, Cardenas Bolivar YR, Montanez Narino V, Stozitzky Rios MV, Arevalo Guerrero CL, Pulido Bobadilla ML, Melo Rojas DM, Lopez Rubio AG, Ortiz Moreno DC, Barreto Garzon PA, Murillo M, Mora-Salamanca AF. Efficacy and safety of the early implementation of a multimodal rehabilitation program in mechanically ventilated patients: A randomized clinical trial protocol. PLoS One. 2025 May 19;20(5):e0324335. doi: 10.1371/journal.pone.0324335. eCollection 2025. PMID 40388519